CLINICAL TRIAL: NCT00746811
Title: A Double-blind, Randomized, Placebo-controlled, Two-period Crossover Trial to Assess the Effects of 4 g/d Prescription Omega-3 Ethyl Esters on Low-density Lipoprotein Cholesterol in Subjects With Primary Hypercholesterolemia
Brief Title: Effects of Prescription Omega-3 on LDL-C in Primary Hypercholesterolemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Provident Clinical Research (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Kevin C. Maki, PhD, Study Director/Chief Science Officer, Provident Clinical Research
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRV-08007
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Primary Hypercholesterolemia
Keywords: cholesterol; hypercholesterolemia; omega 3
MeSH Terms: conditions — Hypercholesterolemia | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- P-OM3 then Placebo (Other): P-OM3 (4 g/d) for the first six weeks of treatment. Placebo (soy oil) for the second six weeks of treatment.
  Interventions: Drug: P-OM3; Drug: Placebo
- Placebo then P-OM3 (Other): Placebo (soy oil) for the first six weeks of treatment. P-OM3 (4 g/d) for the second six weeks of treatment.
  Interventions: Drug: P-OM3; Drug: Placebo

INTERVENTIONS:
Drug: P-OM3 — 4 grams/day - 4 one gram capsules
  Other Names: Lovaza
Drug: Placebo — 4 grams/day - 4 one gram capsules

SUMMARY:
The objectives of this study are to assess the effects of 4 g/d P-OM3, compared with placebo, on LDL-C and other aspects of the fasting lipid profile in subjects with primary hypercholesterolemia.

DETAILED DESCRIPTION:
This trial will utilize a randomized, double-blind, two-period crossover design. At Visit 2 (Week 0), subjects meeting all entry criteria will be randomized to one of two treatment sequences: placebo or P-OM3 for the first 6 week phase followed by the study product they did not receive during the first phase (P-OM3 or placebo) for the second 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18-79 inclusive
* Fasting, untreated low-density lipoprotein cholesterol (LDL-C)level in the borderline high to very high range
* Fasting, untreated triglyceride (TG)level in the normal range
* Provide written informed consent and authorization for protected health information

Exclusion Criteria:

* CHD or CHD risk equivalent
* Pregnancy
* Use of lipid altering medications which cannot be stopped
* Body mass index over 45 kg per square meter
* Allergy or sensitivity to omega-3 fatty acids
* Certain muscle, liver, kidney, lung or gastrointestinal conditions
* Poorly controlled hypertension
* Certain medications
* Active cancers treated within prior 2 years (except non-melanoma skin cancer)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C. Maki, PhD, Study Director — Provident Clinical Research
Locations (1):
- Provident Clinical Research, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Maki KC, Lawless AL, Kelley KM, Dicklin MR, Kaden VN, Schild AL, Rains TM, Marshall JW. Effects of prescription omega-3-acid ethyl esters on fasting lipid profile in subjects with primary hypercholesterolemia. J Cardiovasc Pharmacol. 2011 Apr;57(4):489-94. doi: 10.1097/FJC.0b013e318210fca5. PMID 21297494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted using the research clinic database and print advertisements.
Groups:
- P-OM3 First, Then Placebo: P-OM3 for the first six weeks of treatment. Placebo for the second six weeks of treatment.
  P-OM3: 4 grams/day - 4 one gram capsules
  Placebo: 4 grams/day - 4 one gram capsules
- Placebo First, Then P-OM3: Placebo for the first six weeks of treatment. P-OM3 for the second six weeks of treatment.
  P-OM3: 4 grams/day - 4 one gram capsules
  Placebo: 4 grams/day - 4 one gram capsules
Period: First Intervention (6 Weeks)
Arm/Group | P-OM3 First, Then Placebo | Placebo First, Then P-OM3
Started | 16 | 16
Completed | 15 | 16
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | P-OM3 First, Then Placebo | Placebo First, Then P-OM3
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline/adverse event analyses reported for safety population (all randomized subjects who consumed at least 1 dose of study product; n=31).
Groups:
- Total: Total of all reporting groups
Arm/Group | P-OM3 First, Then Placebo | Placebo First, Then P-OM3 | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (2.1) | 51.2 (2.9) | 54.2 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 27.4 (0.91) | 27.1 (0.85) | 27.3 (0.61)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C During Each Treatment
Description: The primary outcome variable will be the percent change from baseline in LDL-C during each treatment.
  Baseline will be considered the average of values obtained at weeks -1 and 0. On-treatment values will be the average of values collected at weeks 5 and 6 for phase 1, and the average of values collected at weeks 11 and 12 for phase 2.
Time Frame: Baseline (average of weeks -1 and 0) and after 5 or 6 weeks of intervention (average of weeks 5 and 6 for the first treatment phase; average of weeks 11 and 12 for the second treatment phase).
Measure: Mean (Standard Error); unit: Percent change from baseline
Groups:
- P-OM3: P-OM3 for six weeks
  P-OM3: 4 grams/day - 4 one gram capsules
- Placebo: Placebo for six weeks
  Placebo: 4 grams/day - 4 one gram capsules
Arm/Group | P-OM3 | Placebo
Number analyzed (Participants) | 31 | 31
Percent change from baseline | 3.4 (1.8) | -0.7 (1.6)

2. Secondary Outcome: Percent Changes in Other Lipid and Biomarker Levels
Description: Percent changes from baseline in the levels of TC, HDL-C, non-HDL-C, VLDL-C, TG, TC/ HDL-C ratio and Apo AI and B.
  Baseline and on-treatment values for TC, HDL-C, non-HDL-C, VLDL-C, TG, TC/ HDL-C ratio will be calculated as described for LDL-C.
  Baseline values for Apo AI and B will include the average of values obtained at weeks -1 and 0. On-treatment values for Apo AI and B will be the average of values collected at weeks 6 and 12.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change from baseline
Arm/Group | P-OM3 | Placebo
Number analyzed (Participants) | 31 | 31
Percent change from baseline
  TC | 0.5 (1.1) | -0.7 (1.2)
  VLDL-C | -16.7 (3.0) | 2.0 (2.4)
  HDL-C | 1.5 (1.4) | -1.7 (1.2)
  Non-HDL-C | 0.3 (1.6) | -0.4 (1.5)
  TC/HDL-C | -0.6 (1.6) | 1.4 (1.3)
  TG | -16.7 (3.0) | 2.0 (2.4)
  Apo A1 | -2.7 (1.2) | -0.1 (1.2)
  Apo B | -1.2 (1.5) | -1.5 (1.5)

ADVERSE EVENTS:
Groups:
- P-OM3: P-OM3 for the first six weeks of treatment or POM-3 for the second 6 weeks of treatment, depending on group assignment.
  P-OM3: 4 grams/day - 4 one gram capsules
- Placebo: Placebo for the first six weeks of treatment or Placebo for the second 6 weeks of treatment, depending on group assignment.
  Placebo: 4 grams/day - 4 one gram capsules
Arm/Group | P-OM3 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No